CLINICAL TRIAL: NCT04310696
Title: Comparison of Buteyko Breathing Technique and Pursed Lip Breathing to Improve Pulmonary Function in Asthma
Brief Title: Comparison of Buteyko Technique and Pursed Lip Breathing in Asthma
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Riphah International University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: REC/00424 Iqra Arshad Butt
Record Dates: First submitted 2020-03-06; First posted 2020-03-17 (Actual); Last update posted 2020-03-17 (Actual); Status verified 2020-03

CONDITIONS: Asthma
Keywords: Asthma; Buteyko; Pursed lip breathing; Spirometer
MeSH Terms: conditions — Asthma

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Buteyko group (Experimental): Buteyko breathing exercises
  Interventions: Other: Buteyko Breathing exercises
- Pursed lip breathing (Active Comparator): Pursed lip breathing exercises
  Interventions: Other: Pursed lip breathing

INTERVENTIONS:
Other: Buteyko Breathing exercises — Buteyko breathing technique was performed by asking the patient to take a small breath in and then out and hold his/her breath and count the time in seconds, as long as he or she can, until first signs of air hunger start to appear, followed by normal breathing once again. This procedure was repeated 15 times, three sets of 15 repetitions were given to the patient per day, 3 days per week and the treatment was continued for 4 weeks.
  Arms: Buteyko group
Other: Pursed lip breathing — Pursed lip breathing was performed as nasal inspiration followed by expiratory blowing against partially closed lips. Participants received a total of 3 sets of 15 repetitions per day, 3 times a week and the treatment was continued for 4 weeks.
  Arms: Pursed lip breathing

SUMMARY:
The objective of the study was to compare the effects of Buteyko breathing technique and pursed lip breathing technique in the management of asthma. A randomized controlled trial was conducted on 60 asthmatic patients randomly allocated to Buteyko technique group and pursed lip breathing group. Both the groups received 4 weeks of treatment, 3 times per week. Data was collected at base line, 2nd week and 4th week. Outcome measurements included FVC, FEV, PEFR and Asthma Control Test Questionnaire scores. Data analysis was carried out on Statistical Package for the Social Sciences (SPSS) v.21.0. Confidence interval was kept at 95% and a p-value of less than 0.05 was considered significant.

DETAILED DESCRIPTION:
Asthma is an inflammatory condition in which narrowing and swelling of the airways occur, accompanied with extra mucus production. This results in difficulty in breathing and triggers coughing, wheezing and dyspnea. In some cases asthma is a minor irritation, but on the other end of the spectrum it may interfered with activities of daily living and can even become life threatening in severe asthma attacks. According to a study conducted in Pakistan, the prevalence of asthma in adults was found to be 10.8% in adults, working in tanneries with 5.3% of them reporting their symptoms to be work related.

Non-pharmacological management of asthma includes patient education, guidance and physiotherapy. It is suggested that physical therapy may have positive effects in patients with asthma, as they possess dysfunctional breathing patterns accompanied with poor physical condition. Numerous reviews by Cochrane have been published in the recent years regarding the effects of physical therapy in patients with asthma, focusing on the effects of numerous techniques including Alexander technique, manual therapy, physical training, breathing exercises and inspiratory muscle training. In terms of specific effects of different physical therapy treatment techniques in patients with asthma, in light of the existing literature, breathing exercises have found to improve quality of life, reduce symptoms of anxiety, depression and hyperventilation, and decrease respiratory rate and medication use. Moreover, inspiratory muscle training is found to improve symptoms, decrease medication use and also improve inspiratory pressure.

Buteyko technique is a specialized breathing technique developed to reduce chronic hyperinflation.

A pre and post design quasi experimental study conducted was conducted in 2014 to determine the effects of Buteyko breathing technique on asthma control and QOL in school aged children with asthma where Buteyko breathing technique group showed significant improvements terms of asthma control and quality of life.

Based upon the review of the literature, evidence is inadequate in terms of comparison of Buteyko breathing technique with pursed lip breathing technique in the management of patients with asthma except for a single randomized controlled trial. For this reason the purpose of the current study is to compare the effects of Buteyko technique with pursed lip breathing in the management of patients with asthma.

ELIGIBILITY:
Inclusion Criteria:

* Patients categorized as mild to moderate persistent asthma category according to the "National Asthma Education and Prevention Program"

Exclusion Criteria:

* Use of oral steroids within the four-week run-in period,
* Change in inhaled steroid dose and type,
* Other significant unstable medical conditions,
* They have undertaken Buteyko breathing technique previously.

Ages: 18 Years to 40 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 60 (Actual)
Dates: Start 2018-08-30 (Actual); Primary Completion 2019-02-15 (Actual); Study Completion 2019-08-20 (Actual)

PRIMARY OUTCOMES:
Peak expiratory flow rate (PEFR) | After 4 weeks of intervention
  Peak expiratory flow rate (PEFR) measured through digital spirometer. Peak Expiratory Flow Rate (PEFR) measured through digital spirometer. Three zones of measurement are commonly used to interpret peak flow rates. Normal value of PEFR is (80-100%). Green zone indicates 80 to 100 percent of the usual or normal peak flow reading, yellow zone indicates 50 to 79 percent of the usual or normal peak flow readings, and red zone indicates less than 50 percent of the usual or normal peak flow readings.
Forced vital capacity (FVC) | After 4 weeks of intervention
  Forced vital capacity (FVC) measured through digital spirometer. If the value of FVC is within 80% of the reference value, the results are considered normal.
Forced expiratory volume in 1sec (FEV1) | After 4 weeks of intervention
  Forced expiratory volume in 1sec (FEV1) measured through digital spirometer. If the value of FEV1 is within 80% of the reference value, the results are considered normal.
FVC/FEV1 | After 4 weeks of intervention
  FVC/FEV1 measured through digital spirometer. The normal value for the FEV1/FVC ratio is 70% (and 65% in persons older than age 65).
Asthma Control Questionnaire | After 4 weeks of intervention
  Asthma Control questionnaire is a self-reported subjective outcome measurement tool that is used to measure the sufficiency of asthma symptom control and changes in asthma symptoms. It is 5 point scale with scores ranging from 0 to 5 for each item. The greater the score of Asthma Control questionnaire, the better the prognosis and outcome.

CONTACTS AND LOCATIONS:
Overall Officials: Suman Sheraz, PhD*, Principal Investigator — Riphah International University
Locations (1):
- Riphah International University, Islamabad, Federal, Pakistan

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Davies SJ, Jackson PR, Ramsay LE. Dysfunctional breathing and asthma. Panic disorder needs to be considered. BMJ. 2001 Sep 15;323(7313):631; author reply 631-2. No abstract available. PMID 11575318
- [Background] Stoodley I, Williams L, Thompson C, Scott H, Wood L. Evidence for lifestyle interventions in asthma. Breathe (Sheff). 2019 Jun;15(2):e50-e61. doi: 10.1183/20734735.0019-2019. PMID 31777565
- [Background] Arden-Close EJ, Kirby SE, Yardley L, Bruton A, Ainsworth B, Thomas DM. Evaluation of a breathing retraining intervention to improve quality of life in asthma: quantitative process analysis of the BREATHE randomized controlled trial. Clin Rehabil. 2019 Jul;33(7):1139-1149. doi: 10.1177/0269215519832942. Epub 2019 Feb 27. PMID 30813767
- [Background] Singh V, Wisniewski A, Britton J, Tattersfield A. Effect of yoga breathing exercises (pranayama) on airway reactivity in subjects with asthma. Lancet. 1990 Jun 9;335(8702):1381-3. doi: 10.1016/0140-6736(90)91254-8. PMID 1971670
- [Background] Zampogna E, Centis R, Negri S, Fiore E, Cherubino F, Pignatti P, Heffler E, Canonica GW, Sotgiu G, Saderi L, Migliori GB, Spanevello A, Visca D. Effectiveness of pulmonary rehabilitation in severe asthma: a retrospective data analysis. J Asthma. 2020 Dec;57(12):1365-1371. doi: 10.1080/02770903.2019.1646271. Epub 2019 Aug 13. PMID 31317799
- [Background] Austin G. Buteyko technique use to control asthma symptoms. Nurs Times. 2013 Apr 24-30;109(16):16-7. PMID 23697004
- [Background] Barker NJ, Jones M, O'Connell NE, Everard ML. Breathing exercises for dysfunctional breathing/hyperventilation syndrome in children. Cochrane Database Syst Rev. 2013 Dec 18;2013(12):CD010376. doi: 10.1002/14651858.CD010376.pub2. PMID 24347088
- [Background] Wang Q, Zhang W, Liu L, Yang W, Liu H. Effects of physical therapy on lung function in children with asthma: Study protocol for a systematic review and meta-analysis. Medicine (Baltimore). 2019 Apr;98(15):e15226. doi: 10.1097/MD.0000000000015226. PMID 30985726